CLINICAL TRIAL: NCT01081769
Title: A 24-month, Prospective, Randomized, Active-Controlled, Open-Label, Rater-Blinded, Multicenter, International Study of the Prevention of Relapse Comparing Long-Acting Injectable Paliperidone Palmitate to Treatment as Usual With Oral Antipsychotic Monotherapy in Adults With Schizophrenia
Brief Title: Prevention of Relapse With Injectable Paliperidone Palmitate Versus Oral Antipsychotics
Acronym: PROSIPAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015199; R092670SCH3005 (Other: Janssen CTMS ID); 2008-002247-16 (EudraCT Number); NCT01359293 (obsolete NCT alias)
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; paliperidone palmitate; Invega; Intramuscular injection; Oral antipsychotics; Relapse
MeSH Terms: conditions — Schizophrenia; Recurrence | interventions — Paliperidone Palmitate; Antipsychotic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paliperidone Palmitate (Experimental): paliperidone palmitate injection with 150 mg equivalent on Day 1 100 mg equivalent on Day 8 75 mg equivalent on Day 38 and flexible dosing with 25 50 75 100 or 150 mg equivalent once monthly thereafter
  Interventions: Drug: paliperidone palmitate injection
- Oral Antipsychotics (Active Comparator): oral antipsychotics daily treatment according to local label for maximally 24 months
  Interventions: Drug: oral antipsychotics

INTERVENTIONS:
Drug: paliperidone palmitate injection — injection with 150 mg equivalent on Day 1, 100 mg equivalent on Day 8, 75 mg equivalent on Day 38 and flexible dosing with 25, 50, 75, 100 or 150 mg equivalent once monthly thereafter
  Arms: Paliperidone Palmitate
Drug: oral antipsychotics — daily treatment according to local label for maximally 24 months
  Arms: Oral Antipsychotics

SUMMARY:
The purpose of this study is to assess the efficacy (how well the drug works; primarily through the time to relapse) of long-acting injectable paliperidone palmitate compared to treatment as usual with orally administered antipsychotics in monotherapy over 24 months in the treatment of recently diagnosed (1-5 years since diagnosis) schizophrenia.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), open-label (both physician and patient know the name of the assigned drug), rater-blinded (the person who assesses the condition of the patient does not know the name of the assigned drug), active-controlled, parallel-group, multicenter, prospective international study of paliperidone palmitate versus treatment as usual with oral antipsychotic agents in monotherapy in the prevention of relapse (return of symptoms). Patients who have been recently diagnosed with schizophrenia (within 5 years) and are suffering from a schizophrenic relapse (return of symptoms of schizophrenia) will be enrolled. This study consists of a 2-week initial acute oral treatment phase, followed by a treatment phase (core phase) until relapse or up to maximally 24 months, whichever comes first. Prior to a 2-week oral treatment phase, patients will be randomly (by chance) assigned in a 1:1 ratio to receive treatment with paliperidone palmitate injection (once-monthly) or oral antipsychotic medication (daily). Patients randomized to paliperidone palmitate will first receive oral paliperidone ER once daily for 2 weeks followed by paliperidone palmitate injections at a dose of 150 mg eq. on Day 1, 100 mg eq. on Day 8 both in the deltoid muscle and 75 mg eq. on Day 38 and doses in a dose range of 25 to 150 mg eq. in either the deltoid or the gluteal muscle thereafter. Patients randomized to oral comparator arm will receive oral antipsychotics (haloperidol, paliperidone ER, risperidone, olanzapine, quetiapine or aripiprazole) as per investigator discretion and prescribed according to the label. Total treatment duration is maximally 24 months. During the 24 month treatment phase, investigators will be allowed to flexibly decrease or increase the dose of paliperidone palmitate with one dose level in the range of 25 to 150 mg eq. or the oral antipsychotic in the respective locally approved dose range, all according to the patient's clinical needs. The primary endpoint of the 24-month treatment phase will be the time to relapse. Safety will be monitored by evaluating Adverse Events (AEs), rating of extrapyramidal symptoms (symptoms like abnormal muscle movements, abnormal movements of the tongue or jaw, slow or sustained muscle contractions, muscle spasms, shaking, abnormal movements of the eyes, involuntary muscle contractions, slow movements, or restlessness), vital signs measurements (including heart rate and blood pressure), body weight and physical examination findings. A urine pregnancy test will be performed in females of childbearing potential. Adverse events (unintended, but not necessarily unexpected, results of therapy that can be unpleasant or dangerous), associated concomitant medications, and symptoms of relapse will be recorded as needed.

ELIGIBILITY:
Inclusion Criteria:

* Have been meeting the diagnostic criteria for schizophrenia for 1 to 5 years before screening, and have a history of treatment with antipsychotics
* Have a history of two or more relapses requiring psychiatric hospitalization in the preceding 24 months, which may include the current acute episode
* Experiencing at screening an acute schizophrenic episode with a Positive And Negative Syndrome Scale (PANSS) total score at screening between 70 and 120, inclusive
* Be healthy on the basis of physical examination, medical history and vital signs performed at screening
* Woman must be postmenopausal (for at least 1 year) or surgically sterile or abstinent or be practicing an effective method of birth control, must agree to continue to use the same method of contraception throughout the study and must have a negative urine pregnancy test at screening
* be able to fill out questionnaires
* Men must agree to use a double barrier method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study drug

Exclusion Criteria:

* Patients that have never been treated with antipsychotics before
* Treatment resistant patient and/or currently (i.within the last 3 months) treated with clozapine
* Substance dependence within 6 months prior to entry and current intravenous drug use or abuse
* allergies, hypersensitivity, or intolerance to risperidone or paliperidone or excipients
* treatment with a long-acting injectable antipsychotic within three injection cycles prior to screening
* newly started psychotherapy program within the two months preceding the treatment phase baseline
* evidence of clinically significant hepatic, renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances in the past 6 months (as determined by medical history, clinical laboratory or ECG results, or physical examination) that would increase the risk associated with taking study medication or would confound the interpretation of the study
* history or current symptoms of tardive dyskinesia or neuroleptic malignant syndrome
* involuntarily hospitalized patient
* pregnant or breast-feeding females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Start 2010-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (94):
- Vienna, Austria
- Belgium (4):
  - Bertrix
  - Ghent
  - Liège
  - Ostend
- Bulgaria (3):
  - Burgas
  - Plovdiv
  - Radnevo
- Zagreb, Croatia
- Czechia (5):
  - Brno
  - Litoměřice
  - Olomouc
  - Prague
  - Přerov
- Egypt (2):
  - Alexandria
  - Cairo
- Estonia (2):
  - Talinn
  - Tartu
- France (6):
  - Colombes
  - La Seyne-sur-Mer
  - Limoges
  - Metz
  - Paris
  - Saint-Avé
- Germany (4):
  - Berlin
  - Bochum
  - Mannheim
  - München
- Thessalonikis, Greece
- Hungary (4):
  - Budapest
  - Kalocsa
  - Nagykálló
  - Sopron
- Israel (5):
  - Bat Yam
  - Beer Yaakov
  - Hod HaSharon
  - Ramat Gan
  - Tirat Hacarmel
- Amman, Jordan
- Lithuania (2):
  - Šiauliai
  - Vilnius
- Poland (4):
  - Chełmno
  - Gdansk
  - Torun
  - Ząbki
- Romania (5):
  - Arad
  - Bucharest
  - Jebel
  - Oradea
  - Sibiu
- Russia (8):
  - Ekaterinburg Na
  - Krasnodar
  - Nizny Novgorod
  - Saint Petersburg
  - Samara
  - Saratov
  - Tomsk
  - Yaroslavl
- Slovakia (3):
  - Bratislava
  - Michalovce
  - Rimavská Sobota
- South Africa (2):
  - Cape Town
  - Pretoria
- South Korea (4):
  - Goyang
  - Incheon
  - Kyounggi
  - Seoul
- Spain (6):
  - Barcelona
  - Burgos
  - Elche
  - Madrid
  - Sant Boi de Llobregat
  - Zamora
- Taiwan (3):
  - Taichung
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (3):
  - Istanbul
  - Manisa Turkey
  - Zonguldak
- Ukraine (11):
  - Dnipropetrovsk
  - Donetsk
  - Hlevakha
  - Kharkiv
  - Kherson
  - Kiev
  - Lviv
  - Odesa
  - Poltava
  - Simferopol
  - Uzhhorod
- United Kingdom (4):
  - Birmingham
  - Exeter
  - London
  - Warrington

REFERENCES:
- [Derived] Lopena OJ, Alphs LD, Sajatovic M, Turkoz I, Sun L, Johnston KL, Sliwa JK, Najarian DM, Starr HL. Earlier Use of Long-Acting Injectable Paliperidone Palmitate Versus Oral Antipsychotics in Patients With Schizophrenia: An Integrated Patient-Level Post Hoc Analysis. J Clin Psychiatry. 2023 Sep 25;84(6):23m14788. doi: 10.4088/JCP.23m14788. PMID 37756123

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After randomization patients enrolled in a 2-week oral treatment phase and were considered part of the whole Intent-to-Treat population (Whole ITT). Five patients did not receive study medication after randomization and were excluded from the whole ITT. Only responders were considered for continuation in the Core treatment phase (Core ITT).
Groups:
- Paliperidone Palmitate: 2 weeks oral paliperidone treatment followed by intramuscular injection with 150 mg paliperidone palmitate equivalent on Day 1 of the core treatment phase, 100 mg equivalent on Day 8, 75 mg equivalent on Day 38 and flexible dosing with 25, 50, 75, 100 or 150 mg equivalent once monthly thereafter
Period: Whole Intent-to-Treat
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Started | 376 | 388
Completed | 352 | 363
Not Completed | 24 | 25
Not completed — Missing Responder Assessment | 10 | 12
Not completed — Stopped; non-responder after 2 weeks | 6 | 6
Not completed — Deviation; non-responder after 2 weeks | 6 | 7
Not completed — Responder after 2 weeks, but stopped | 2 | 0
Period: CORE Intent-To-Treat
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Started | 352 | 363
Completed | 272 | 266
Not Completed | 80 | 97
Not completed — Adverse Event | 14 | 11
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 2 | 6
Not completed — Lost to Follow-up | 4 | 5
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 52 | 60
Not completed — Noncompliance With Study Drug | 0 | 5
Not completed — Other | 0 | 1
Not completed — Ineligibility | 3 | 4
Not completed — Visit Schedule Issues | 1 | 2
Not completed — Patient Moved | 2 | 2

BASELINE CHARACTERISTICS:
Population: Whole Intent-to-Treat population: All randomized patients who received at least 1 dose of study medication during the screening or treatment phase
Groups:
- Total: Total of all reporting groups
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics | Total
Number analyzed (Participants) | 376 | 388 | 764
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (10.73) | 32.4 (10) | 32.5 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 171 | 318
  Male | 229 | 217 | 446
Region of Enrollment [Number; unit: participants]
  AUSTRIA | 0 | 1 | 1
  BELGIUM | 7 | 5 | 12
  BULGARIA | 15 | 15 | 30
  CROATIA | 12 | 12 | 24
  CZECH REPUBLIC | 14 | 21 | 35
  EGYPT | 16 | 14 | 30
  ESTONIA | 2 | 3 | 5
  FRANCE | 4 | 4 | 8
  GERMANY | 3 | 2 | 5
  HUNGARY | 15 | 16 | 31
  ISRAEL | 6 | 5 | 11
  ITALY | 10 | 11 | 21
  JORDAN | 15 | 11 | 26
  KOREA, REPUBLIC OF KOREA | 2 | 4 | 6
  LITHUANIA | 13 | 14 | 27
  POLAND | 11 | 11 | 22
  ROMANIA | 13 | 14 | 27
  RUSSIAN FEDERATION | 90 | 90 | 180
  SLOVAKIA | 13 | 14 | 27
  SOUTH AFRICA | 26 | 24 | 50
  SPAIN | 3 | 4 | 7
  TAIWAN, PROVINCE OF CHINA | 4 | 5 | 9
  TURKEY | 11 | 9 | 20
  UKRAINE | 71 | 79 | 150

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse Event
Description: Number of days from baseline (day 1 of core phase) to relapse as evaluated according the Csernansky criteria. A patient was considered to have relapsed if they met one or more of the following criteria: (1) psychiatric hospitalization; (2) an increase in the level of psychiatric care and an increase of 25 percent (%) from baseline in the Positive And Negative Syndrome Score (PANSS) total score (or an increase of 10 points if the baseline score was 40 or less); (3) deliberate self-injury; (4) suicidal or homicidal ideation that was clinically significant in the investigator's judgment; (5) violent behavior resulting in clinically significant injury to another person or property damage; (6) substantial clinical deterioration, defined as a change score of 6 ("much worse") or 7 ("very much worse") on the Clinical Global Impressions Scale (CGI-C); and/or (7) the required dose of the antipsychotic exceeds the maximum approved dose.
Time Frame: from baseline (Day 1 of core phase) up to maximally 24 months.
Population: all randomized subjects who responded at the end of the 2-week initial acute oral treatment phase, who also received at least one dose of study medication during the 24-month core treatment phase and provided at least one post-baseline efficacy assessment
Measure: Mean (Standard Error); unit: days
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
days | 616 (10.9) | 603 (13.1)
Statistical Analysis 1: Comparison: Paliperidone Palmitate vs Oral Antipsychotics; Test type: Superiority or Other; p = 0.0191, Log Rank

2. Secondary Outcome: Percentage of Treatment Responders
Description: The proportion of patients achieving a treatment response, defined as a ≥30% decrease (i.e., improvement) in Positive and Negative Syndrome Scale (PANSS) total score from baseline to endpoint. The PANSS is a 30-item scale (Range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate increased severity of schizophrenia symptoms.
Time Frame: from baseline (day 1 of core phase) up to maximally 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
percentage of participants | 75.6 [70.8 to 79.8] | 69.4 [64.5 to 73.9]

3. Secondary Outcome: Change From Baseline in PANSS Total Score
Description: Change from baseline in the PANSS: The PANSS is a 30-item scale (Range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate worsening.
Time Frame: Baseline, day 8, month 1, 2, 3, 4, 6, 9, 12, 15, 18, 21, 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
units on a scale
  Baseline score | 82.5 (12.03) | 81.5 (11.70)
  change from baseline at Day 8 | -4.8 (5.93) | -3.7 (7.04)
  change from baseline at Month 1 | -9.4 (10.91) | -8.8 (10.15)
  change from baseline at Month 2 | -12.2 (12.19) | -12.3 (11.34)
  change from baseline at Month 3 | -14.5 (11.72) | -15.0 (11.15)
  change from baseline at Month 4 | -16.2 (13.03) | -16.8 (12.34)
  change from baseline at Month 6 | -18.5 (13.67) | -18.6 (13.09)
  change from baseline at Month 9 | -19.5 (14.72) | -20.1 (14.35)
  change from baseline at Month 12 | -21.8 (13.32) | -21.2 (14.45)
  change from baseline at Month 15 | -21.7 (14.56) | -21.9 (14.18)
  change from baseline at Month 18 | -23.5 (13.56) | -22.8 (14.41)
  change from baseline at Month 21 | -24.3 (13.60) | -23.7 (14.66)
  change from baseline at Month 24 | -25.5 (14.42) | -24.6 (14.16)
  change at Endpoint (LOCF) | -16.6 (21.42) | -14.1 (21.29)

4. Secondary Outcome: Change From Baseline in PANSS Subscale Score
Description: Change from baseline in positive symptom, negative symptom and general psychopathology subscales of the PANSS scale. The PANSS scale is designed to assess symptoms of schizophrenia by means of the 30-items. The PANSS scale provides subscores for 3 subscales, that is, the positive symptoms subscale (7 items, range 7-49), the negative symptoms subscale (7 items, range 7-49), and the general psychopathology subscale (16 items, range 16-112). Each item of the scale is to be scored on a scale of 1 (absent) to 7 (extreme). Higher scores indicate higher severity of schizophrenia symptoms.
Time Frame: Baseline (day 1 of core phase), day 8, month 12, 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
units on a scale
  Positive Subscale; Baseline score | 18.4 (3.97) | 18.3 (4.01)
  Positive Subscale; change at Day 8 | -1.5 (2.11) | -1.3 (2.36)
  Positive Subscale; change at Month 12 | -6.3 (4.10) | -6.2 (4.35)
  Positive Subscale; change at Month 24 | -6.8 (4.39) | -6.7 (4.48)
  Positive Subscale; change at Endpoint (LOCF) | -4.4 (6.61) | -3.8 (6.72)
  Negative Subscale; Baseline score | 22.6 (4.55) | 22.3 (4.58)
  Negative Subscale; change at Day 8 | -1.0 (1.90) | -0.8 (2.10)
  Negative Subscale; change at Month 12 | -4.8 (4.69) | -4.7 (4.80)
  Negative Subscale; change at Month 24 | -6.2 (5.19) | -5.9 (4.74)
  Negative Subscale; change at Endpoint (LOCF) | -4.1 (6.13) | -3.7 (5.79)
  General Psychopathology; Baseline score | 41.4 (6.73) | 40.8 (6.59)
  General Psychopathology; change at Day 8 | -2.3 (3.58) | -1.6 (4.01)
  General Psychopathology; change at Month 12 | -10.7 (7.19) | -10.3 (7.64)
  General Psychopathology; change at Month 24 | -12.5 (7.63) | -12.0 (7.82)
  General Psychopathology; change at Endpoint (LOCF) | -8.1 (10.96) | -6.7 (11.12)

5. Secondary Outcome: Change From Baseline in PANSS Marder Factor Scores
Description: Change from baseline in schizophrenia symptoms were assessed through the following PANSS factor scores as described by Marder: (1) positive symptoms (range 8-56): sum of delusions, hallucinatory behavior, grandiosity, suspiciousness, stereotyped thinking, somatic concern, unusual thought content, lack of judgment and insight; (2) negative symptoms (range 7-49): sum of blunted affect, emotional withdrawal, poor rapport, passive social withdrawal, lack of spontaneity, motor retardation, and active social avoidance; (3) disorganized thoughts (range 7-49): sum of conceptual disorganization, difficulty in abstract thinking, mannerisms and posturing, disorientation, poor attention, disturbance of volition, and preoccupation; (4) uncontrolled hostility/excitement (range 4-28): sum of excitement, hostility, uncooperativeness and poor impulse control; (5) anxiety/depression (range 4-28): sum of anxiety, guilt feelings, tension, and depression. Higher scores indicate higher severity of symptoms
Time Frame: Baseline (day 1 of core phase), day 8, month 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
units on a scale
  Positive Symptoms Factor Score; Baseline score | 22.9 (4.26) | 22.5 (4.39)
  Positive Symptoms Factor Score; change at Day 8 | -1.5 (2.22) | -1.3 (2.50)
  Positive Symptoms Factor Score; change at Month 12 | -6.9 (4.31) | -6.9 (4.76)
  Positive Symptoms Factor Score; change at Month 24 | -7.6 (4.48) | -7.8 (4.95)
  Positive Symptoms Factor Score; change at Endpoint | -5.0 (6.73) | -4.7 (6.80)
  Negative Symptoms Factor Score; Baseline score | 22.0 (4.65) | 21.5 (4.95)
  Negative Symptoms Factor Score; change at Day 8 | -1.0 (1.93) | -0.8 (2.25)
  Negative Symptoms Factor Score; change at Month 12 | -5.1 (4.73) | -4.9 (4.88)
  Negative Symptoms Factor Score; change at Month 24 | -6.5 (5.16) | -6.1 (5.05)
  Negative Symptoms Factor Score; change at Endpoint | -4.3 (6.26) | -3.8 (6.08)
  Disorganized Thoughts Factor; Baseline score | 19.5 (3.54) | 19.4 (3.41)
  Disorganized Thoughts Factor; change at Day 8 | -1.0 (1.61) | -0.6 (2.06)
  Disorganized Thoughts Factor; change at Month 12 | -4.6 (3.42) | -4.6 (3.78)
  Disorganized Thoughts Factor; change at Month 24 | -5.4 (3.90) | -5.4 (3.82)
  Disorganized Thoughts Factor; change at Endpoint | -3.7 (5.03) | -3.2 (5.16)
  Uncontrolled Hostility/Excitement; Baseline score | 8.4 (2.71) | 8.3 (2.64)
  Uncontrolled Hostility/Excitement; change at Day 8 | -0.7 (1.60) | -0.4 (1.47)
  Uncontrolled Hostility/Excitement; change Month 12 | -2.3 (2.57) | -2.1 (2.62)
  Uncontrolled Hostility/Excitement; change Month 24 | -2.7 (2.77) | -2.3 (2.73)
  Uncontrolled Hostility/Excitement; change Endpoint | -1.5 (3.82) | -0.8 (3.87)
  Anxiety/Depression Factor; Baseline score | 9.7 (2.74) | 9.8 (2.85)
  Anxiety/Depression Factor; change at Day 8 | -0.8 (1.57) | -0.6 (1.72)
  Anxiety/Depression Factor; change at Month 12 | -2.8 (2.67) | -2.7 (2.56)
  Anxiety/Depression Factor; change at Month 24 | -3.3 (2.90) | -3.0 (2.78)
  Anxiety/Depression Factor; change at Endpoint | -2.1 (3.51) | -1.8 (3.47)

6. Secondary Outcome: Change From Baseline in Clinical Global Impression Severity (CGI-S) Score
Description: The Clinical Global Impression Severity (CGI-S) rating scale is a 7 point global clinical assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate higher impression of illness severity.
Time Frame: Baseline (day 1 of core phase), day 8, month 1, 2, 3, 4, 6, 9, 12, 15, 18, 21, 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
units on a scale
  Baseline score | 3.9 (0.37) | 3.8 (0.40)
  change from baseline at Day 8 | -0.1 (0.38) | -0.1 (0.43)
  change from baseline at Month 1 | -0.3 (0.61) | -0.3 (0.61)
  change from baseline at Month 2 | -0.4 (0.70) | -0.5 (0.71)
  change from baseline at Month 3 | -0.6 (0.69) | -0.6 (0.69)
  change from baseline at Month 4 | -0.7 (0.75) | -0.8 (0.71)
  change from baseline at Month 6 | -0.8 (0.78) | -0.8 (0.73)
  change from baseline at Month 9 | -0.9 (0.80) | -0.9 (0.78)
  change from baseline at Month 12 | -1.0 (0.78) | -1.0 (0.80)
  change from baseline at Month 15 | -0.9 (0.82) | -1.0 (0.80)
  change from baseline at Month 18 | -1.0 (0.80) | -1.0 (0.78)
  change from baseline at Month 21 | -1.0 (0.78) | -1.1 (0.82)
  change from baseline at Month 24 | -1.1 (0.79) | -1.1 (0.80)
  change from baseline at Endpoint (LOCF) | -0.7 (1.14) | -0.6 (1.12)

7. Secondary Outcome: Clinical Global Impression-Change (CGI-C)
Description: The Clinical Global Impression-Change (CGI-C) rating scale is used to rate the change in severity of the patient's illness compared to baseline (day 1 of core phase) on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Month 24 and endpoint
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
percentage of participants
  Month 24; Very Much Improved | 22.9 (22.9) | 21.7 (21.7)
  Month 24; Much Improved | 52.9 (52.9) | 47.8 (47.8)
  Month 24; Minimally Improved | 17.0 (17.0) | 20.8 (20.8)
  Month 24; No change | 6.7 (6.7) | 7.7 (7.7)
  Month 24; Minimally Worse | 0.0 (0.0) | 1.0 (1.0)
  Month 24; Much Worse | 0.4 (0.4) | 1.0 (1.0)
  Month 24; Very Much Worse | 0.0 (0.0) | 0.0 (0.0)
  Endpoint; Very Much Improved | 17.1 (17.1) | 14.2 (14.2)
  Endpoint; Much Improved | 40.6 (40.6) | 35.8 (35.8)
  Endpoint; Minimally Improved | 17.4 (17.4) | 21.9 (21.9)
  Endpoint; No change | 10.6 (10.6) | 10.8 (10.8)
  Endpoint; Minimally Worse | 5.1 (5.1) | 6.1 (6.1)
  Endpoint; Much Worse | 9.1 (9.1) | 10.6 (10.6)
  Endpoint; Very Much Worse | 0.0 (0.0) | 0.6 (0.6)

8. Secondary Outcome: Changes From Baseline in Personal and Social Performance (PSP) Total Score
Description: The Personal and Social Performance (PSP) scale assesses degree of a participant's dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. Score ranges from 1 to 100, divided into 10 equal intervals to rate degree of difficulty (1, absent to 6, very severe) in each of the 4 domains. Based on 4 domains there will be 1 total score. Participants with score of 71 to 100 have mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision.
Time Frame: baseline (day 1 of core phase), month 1, 3, 6, 9, 12, 15, 18, 21 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
units on a scale
  Baseline score | 55.3 (11.31) | 55.3 (11.07)
  change from baseline at Month 1 | 4.9 (7.78) | 4.3 (7.65)
  change from baseline at Month 3 | 7.6 (8.91) | 7.7 (9.02)
  change from baseline at Month 6 | 9.9 (10.08) | 10.8 (10.32)
  change from baseline at Month 9 | 11.4 (11.28) | 11.9 (11.03)
  change from baseline at Month 12 | 12.7 (10.78) | 12.3 (11.27)
  change from baseline at Month 15 | 12.9 (11.05) | 12.9 (10.82)
  change from baseline at Month 18 | 14.0 (11.44) | 13.3 (11.44)
  change from baseline at Month 21 | 14.7 (12.3) | 14.0 (11.69)
  change from baseline at Month 24 | 15.2 (12.72) | 14.6 (11.72)
  change from baseline at Endpoint (LOCF) | 9.8 (15.41) | 8.7 (14.89)

9. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36)
Description: The Short Form-36 Health Survey (SF-36) is a measure of Participant-reported health status. It is a 36-item questionnaire measuring 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health). Two summary scale scores are computed based on weighted combinations of the 8 subscale scores: the Physical Component Summary and the Mental Component Summary. Each summary scale score ranges from 0 (worst) to 100 (best), with higher scores reflecting better health-related functional status.
Time Frame: baseline (day 1 of core phase), month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
units on a scale
  Physical Component, Baseline score | 50.3 (8.04) | 50.6 (7.83)
  Physical Component, change at Month 6 | 1.2 (6.92) | 1.3 (6.52)
  Physical Component, change at Month 12 | 1.6 (7.62) | 1.2 (7.08)
  Physical Component, change at Month 24 | 2.2 (8.40) | 2.1 (6.74)
  Physical Component, change at Endpoint (LOCF) | 1.7 (8.52) | 1.4 (7.40)
  Mental Component, Baseline score | 32.1 (12.62) | 31.4 (12.92)
  Mental Component, change at Month 6 | 8.2 (11.58) | 9.1 (12.43)
  Mental Component, change at Month 12 | 10.5 (11.75) | 11.6 (12.77)
  Mental Component, change at Month 24 | 12.0 (13.34) | 12.3 (12.83)
  Mental Component, change at Endpoint (LOCF) | 9.0 (14.99) | 8.7 (14.37)

10. Secondary Outcome: Change From Baseline in EuroQol 5-Dimensional Questionnaire (EQ-5D) VAS Score
Description: The EQ-5D VAS records the respondent's self-rated health on a vertical, visual analog scale, with 0 representing the worst imaginable health state and 100 representing the best imaginable health state. The EQ VAS is used as a quantitative measure of health outcome as judged by the individual respondent.
Time Frame: baseline (day 1 of core phase), month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
units on a scale
  Baseline score | 57.5 (20.94) | 57.6 (20.41)
  change from baseline at Month 6 | 10.6 (17.31) | 11.9 (17.00)
  change from baseline at Month 12 | 15.0 (17.38) | 15.6 (18.32)
  change from baseline at Month 24 | 17.9 (19.48) | 18.6 (17.36)
  change from baseline at Endpoint (LOCF) | 13.0 (22.87) | 11.9 (21.54)

11. Secondary Outcome: Change From Baseline in EuroQol 5-Dimensional Questionnaire (EQ-5D) Index Score
Description: The EuroQol-5 is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead. A higher score indicates an improvement in health in the Health Status Index.
Time Frame: baseline (day 1 of core phase), month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
units on a scale
  Baseline score | 0.80 (0.173) | 0.78 (0.181)
  change from baseline at Month 6 | 0.06 (0.181) | 0.09 (0.157)
  change from baseline at Month 12 | 0.08 (0.185) | 0.11 (0.179)
  change from baseline at Month 24 | 0.10 (0.201) | 0.12 (0.161)
  change from baseline at Endpoint (LOCF) | 0.06 (0.224) | 0.08 (0.192)

12. Secondary Outcome: Change From Baseline in Subjective Well-Being Under Neuroleptics-Short Form (SWN-S) Total Score
Description: The SWN-S is a patient self-rated scale developed to measure the subjective well-being for the previous 7 days of a patient under neuroleptic treatment. The SWN-S consists of 20 items (each item is rated from 1=not at all to 6=very much). The total score ranges from 20 to 120 with higher score indicating greater subjective well-being.
Time Frame: baseline (day 1 of core phase), month 6, 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
units on a scale
  Baseline score | 76.5 (17.02) | 76.7 (17.07)
  change from baseline at Month 6 | 8.4 (14.06) | 9.1 (14.40)
  change from baseline at Month 12 | 11.4 (15.81) | 11.1 (17.02)
  change from baseline at Month 24 | 13.4 (18.14) | 13.1 (15.76)
  change from baseline at Endpoint (LOCF) | 9.7 (19.17) | 8.3 (17.58)

13. Secondary Outcome: Change From Baseline in Patient's Treatment Satisfaction
Description: Patient's satisfaction with medication was assessed using the Treatment Satisfaction Questionnaire for Medication (TSQM). The TSQM is divided into 4 subscales (effectiveness, side effects, convenience, and global satisfaction), with the value of each subscale ranging from 0 to 100. Higher scores indicate greater treatment satisfaction.
Time Frame: baseline (day 1 of core phase), month 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
units on a scale
  Effectiveness; Baseline score | 61.9 (16.97) | 59.5 (16.82)
  Effectiveness; change at Month 12 | 6.7 (22.72) | 6.6 (21.99)
  Effectiveness; change at Month 24 | 8.5 (21.75) | 12.4 (20.69)
  Effectiveness; change at Endpoint (LOCF) | 3.8 (23.47) | 4.5 (25.31)
  Side-effects; Baseline score | 91.3 (19.74) | 87.3 (23.41)
  Side-effects; change at Month 12 | 2.1 (22.71) | 2.5 (25.66)
  Side-effects; change at Month 24 | 2.8 (20.93) | 3.5 (23.96)
  Side-effects; change at Endpoint (LOCF) | -1.4 (25.59) | 0.7 (28.24)
  Convenience; Baseline score | 67.1 (16.66) | 68.4 (16.45)
  Convenience; change at Month 12 | 8.4 (19.10) | 1.0 (17.79)
  Convenience; change at Month 24 | 10.4 (20.49) | 4.7 (17.69)
  Convenience; change at Endpoint (LOCF) | 7.4 (21.24) | 0.3 (21.68)
  Global Satisfaction; Baseline score | 64.0 (18.13) | 62.8 (18.31)
  Global Satisfaction; change at Month 12 | 8.2 (18.89) | 7.0 (21.18)
  Global Satisfaction; change at Month 24 | 8.6 (21.06) | 9.2 (20.39)
  Global Satisfaction; change at Endpoint (LOCF) | 3.0 (25.01) | 1.0 (26.76)

14. Secondary Outcome: Change From Baseline in Physician's Treatment Satisfaction
Description: Physician's treatment satisfaction was assessed using the physician's treatment satisfaction scale which is designed to rate 4 aspects of treatment (efficacy, safety, mode of administration, and overall satisfaction), each on a scale ranging from 1 (extremely satisfied) to 7 (extremely dissatisfied).
Time Frame: baseline (day 1 of core phase), month 12 and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
units on a scale
  Efficacy; Baseline score | 2.7 (0.79) | 2.8 (0.79)
  Efficacy; change at Month 12 | -0.5 (1.03) | -0.4 (0.92)
  Efficacy; change at Month 24 | -0.6 (1.10) | -0.6 (0.98)
  Efficacy; change at Endpoint (LOCF) | -0.2 (1.46) | 0.0 (1.43)
  Safety; Baseline score | 2.4 (0.80) | 2.6 (0.77)
  Safety; change at Month 12 | -0.4 (0.97) | -0.2 (0.90)
  Safety; change at Month 24 | -0.4 (0.97) | -0.3 (1.04)
  Safety; change at Endpoint (LOCF) | -0.2 (1.19) | -0.0 (1.18)
  Mode of Administration: Baseline score | 2.6 (0.86) | 2.6 (0.83)
  Mode of Administration: change at Month 12 | -0.7 (1.02) | -0.0 (0.92)
  Mode of Administration: change at Month 24 | -0.7 (1.09) | -0.1 (0.92)
  Mode of Administration: change at Endpoint (LOCF) | -0.5 (1.16) | 0.0 (1.04)
  Overall Satisfaction; Baseline score | 2.6 (0.78) | 2.7 (0.74)
  Overall Satisfaction; change at Month 12 | -0.5 (0.95) | -0.3 (0.84)
  Overall Satisfaction; change at Month 24 | -0.6 (1.00) | -0.3 (0.86)
  Overall Satisfaction; change at Endpoint (LOCF) | -0.2 (1.25) | 0.1 (1.16)

15. Primary Outcome: Number of Participants With a Relapse Event
Description: Number of participants with a relapse event with relapses evaluated according the Csernansky criteria. A patient was considered to have relapsed if they met one or more of the following criteria: (1) psychiatric hospitalization; (2) an increase in the level of psychiatric care and an increase of 25% from baseline in the PANSS total score (or an increase of 10 points if the baseline score was 40 or less); (3) deliberate self-injury; (4) suicidal or homicidal ideation that was clinically significant in the investigator's judgment; (5) violent behavior resulting in clinically significant injury to another person or property damage; (6) substantial clinical deterioration, defined as a change score of 6 ("much worse") or 7 ("very much worse") on the Clinical Global Impressions Scale (CGI-C); and/or (7) the required dose of the antipsychotic exceeds the maximum approved dose.
Time Frame: from baseline (Day 1 of core phase) up to maximally 24 months
Population: as for outcome 1
Measure: Number; unit: number of participants
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 352 | 363
number of participants
  No | 300 | 287
  Yes | 52 | 76
Statistical Analysis 1: Comparison: Paliperidone Palmitate vs Oral Antipsychotics; Test type: Superiority or Other; p = 0.0323, Fisher Exact

ADVERSE EVENTS:
Time Frame: from randomization until maximally month 24
Description: Only patients who had at least one of the TEAEs listed in the Other (non Serious) AE table are included in the Total no. subjects with Non-Serious Adverse Events
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Serious Adverse Events (participants affected / at risk) | 42/376 | 48/388
Other Adverse Events (participants affected / at risk) | 208/376 | 208/388
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Palmitate (N=376) | Oral Antipsychotics (N=388)
Cardiac arrest (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Hepatic echinococciasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Prognathism (Musculoskeletal and connective tissue disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Acute psychosis (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 2
Alcohol abuse (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 0
Psychotic disorder (Psychiatric disorders) | 7 | 8
Schizophrenia (Psychiatric disorders) | 21 | 22
Schizophrenia, paranoid type (Psychiatric disorders) | 3 | 4
Suicide attempt (Psychiatric disorders) | 0 | 2
Calculus bladder (Renal and urinary disorders) | 1 | 0
Varicocele (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Palmitate (N=376) | Oral Antipsychotics (N=388)
Vertigo (Ear and labyrinth disorders) | 8 | 6
Diarrhoea (Gastrointestinal disorders) | 8 | 7
Nausea (Gastrointestinal disorders) | 12 | 13
Asthenia (General disorders) | 7 | 8
Fatigue (General disorders) | 9 | 7
Injection site pain (General disorders) | 24 | 0
Influenza (Infections and infestations) | 6 | 8
Nasopharyngitis (Infections and infestations) | 25 | 20
Weight decreased (Investigations) | 9 | 9
Weight increased (Investigations) | 58 | 65
Increased appetite (Metabolism and nutrition disorders) | 9 | 12
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 12 | 8
Akathisia (Nervous system disorders) | 21 | 22
Headache (Nervous system disorders) | 40 | 34
Sedation (Nervous system disorders) | 6 | 10
Somnolence (Nervous system disorders) | 13 | 22
Tremor (Nervous system disorders) | 22 | 17
Agitation (Psychiatric disorders) | 9 | 9
Anxiety (Psychiatric disorders) | 22 | 23
Depression (Psychiatric disorders) | 11 | 9
Insomnia (Psychiatric disorders) | 42 | 39
Schizophrenia (Psychiatric disorders) | 9 | 15
Suicidal ideation (Psychiatric disorders) | 20 | 23
Amenorrhoea (Reproductive system and breast disorders) | 11 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the Sponsor for review at least 60 days prior to submission for publication or presentation.

No paper that incorporates Confidential Information will be submitted for publication without Sponsor's prior written consent. If requested in writing, such publication will be withheld for up to an additional 60 calendar days. A publication from the individual Study site data will not be published until the combined results have been published.